CLINICAL TRIAL: NCT00592865
Title: Genetic Epidemiology of Adult Brain Tumors
Brief Title: Risk Factors for Adult-Onset Brain Tumors
Status: Terminated | Type: Observational
Sponsor: Vanderbilt University Medical Center (Other)
Collaborators: H. Lee Moffitt Cancer Center and Research Institute (Other); Kentuckiana Cancer Institute (Other); Emory University (Other); University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Reid Thompson, Department Chair and Professor, Neurological Surgery, Vanderbilt University Medical Center
Other Study IDs: 030917
Record Dates: First submitted 2008-01-07; First posted 2008-01-14 (Estimated); Last update posted 2021-02-21 (Actual); Status verified 2021-02

CONDITIONS: Brain Neoplasm, Primary; Brain Neoplasms, Malignant; Brain Neoplasms, Benign
MeSH Terms: conditions — Brain Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Biospecimen Retention: Samples With DNA — Mouthwash and salvia samples. Toenail samples are also collected.
Oversight: Data Monitoring Committee: No

SUMMARY:
Study Objective:

Brain tumors are poorly understood. The purpose of this research is to examine whether factors in lifestyle play a role in brain tumor development. The study will also investigate the contribution of inherited susceptibility to the risk of brain cancer. By gaining a better understanding of these influences, the investigators hope to learn how to prevent brain tumors in future generations, and to develop more effective strategies for treatment.

Study Protocol:

This is a case-control investigation. Persons affected with a brain tumor are compared to unaffected persons on previous medical history, diet and other factors. Those enrolled in the study will participate in an interview on general background, diet, medical history and lifestyle, and will provide a sample of DNA, clippings of your toenails, and a tap water sample from your home. All procedures are performed in the clinic or through the mail.

'Cases': Cases eligible for the study are persons with a recent diagnosis of a primary brain tumor (glioma or meningioma), at least 18 years of age.

'Controls': Controls in the study are non-family members of patients, similar in age and of the same gender. Suitable controls include in-laws, friends, neighbors and co-workers.

DETAILED DESCRIPTION:
Primary Objective:

The primary objective of this research is to establish a clinic-based case-control study for examination of potential risk factors for primary adult brain tumors. After assembling a series of 1,500 cases and 3,000 controls, investigators will test current hypotheses on ge-netic and environmental risk factors for the occurrence of these tumors.

STUDY DESIGN:

In this case-control study, persons with a recent diagnosis (within 4 months) of a primary brain tumor will be identified in the neurology/neurosurgery clinics at major treatment referral centers in the Southeast. Non-blood related relatives (eg. in-laws), friends or other persons will be recruited as controls. Names and contact information of eligible controls will be ascertained from patients. A total of 1,500 cases and 3,000 controls will be enrolled over the course of the 5-year study. All enrolled subjects will complete a one hour interview on lifestyle, environmental exposures, diet, physical activity, tobacco use and medical history. They will also be asked to provide a DNA sample, a water sample and a toenail sample (from each great toe). At the end of data collection, lifestyles and genetic attributes will be compared in cases and controls to identify any differences that may be relevant to the causation of disease. Because the study will recruit patients near the time of disease diagnosis, full enrollment should be possible. In addition, high re-sponse rates are anticipated among the controls. Thus, with the large numbers of patients available and high anticipated response rates, the study offers a unique opportunity to successfully identify environmental and genetic risk factors for this uncommon form of cancer.

ELIGIBILITY:
Inclusion Criteria:

* Case: Incident primary glioma or meningioma of any stage, diagnosed within 4 months.
* Control: non-blood relative, friend, co-worker of same gender as case
* Aged 18 and older; either gender; any race

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: "Case" subjects will be identified from the patients referred to neurology/neurosurgery clinics. Cases, when enrolled in the study, will be asked to identify potential "controls" by providing the name and phone number of the same-sex in-law nearest in age to the case and/or the name of a same-sex friend will also be sought.
Sampling Method: Non-Probability Sample
Enrollment: 850 (Actual)
Dates: Start 2003-10; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kathleen M. Egan, DSc, Principal Investigator — H. Lee Moffitt Cancer Center; Reid C. Thompson, MD, Principal Investigator — Vanderbilt University Medical Center; Renato V. LaRocca, MD, Principal Investigator — Kentuckiana Cancer Center; Jeffrey Olson, MD, Principal Investigator — Emory University; Burt Nabors, MD, Principal Investigator — University of Alabama at Birmingham
Locations (5):
- United States (5):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - H. Lee Moffitt Cancer Center, Tampa, Florida
  - Emory University, Atlanta, Georgia
  - Kentuckaina Cancer Institute, Louisville, Kentucky
  - Vanderbilt University Medical Center, Department of Neurological Surgery, Nashville, Tennessee

IPD SHARING:
Plan to Share IPD: No